CLINICAL TRIAL: NCT04879667
Title: Endoscopic Management Of Refractory Gastro-cutaneous Fistula After Laparoscopic Sleeve Gastrectomy ; A Randomized Control Trial
Brief Title: Endoscopic Management Of Refractory Gastro-cutaneous Fistula After Laparoscopic Sleeve Gastrectomy l
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Said Mohamed Said Abdou Negm, lecturer of general surgery, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zagazig University Hospitalis
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Bariatric Surgery Candidate
Keywords: Laparoscopic Sleeve Gastrectomy

STUDY DESIGN:
Intervention Model Description: This study included patients who were admitted to investigators' center to do laparoscopic sleeve gastrectomy and complicated by gastro-cutaneous fistula . Cases were collected in the period from December 2019 to march 2021. the sample size was 30 patients divided into two equal groups. Group (1) included 15 patients managed by surgical intervention , group (2) included 15 patients managed by endoscopic intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (1) (No Intervention): surgical management of gastrocutaneous fistula after laparoscopic sleeve gatrectomy by surgical exploration
- group (2) (Active Comparator): we performed upper GI endoscopy to all cases first to assess the site , size and cause of fistula . we used stents , clips , sutures and ballon dilatation to close the fistula according to size , site and cause of fistula.if the fistula had no track that was proved by CT with oral & I.V contrast , we used the endoscopic stent. if the fistula had track that was proved by CT with oral & I.V contrast , we used the OVASCO clip , endo suturing or ballon. Combined maneuvers may be used like ballon dilation and clipping or ballon dilatation and suturing if there was distal narrowing.
  Interventions: Procedure: endoscopic management of gastrocutaneous fistula after laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: endoscopic management of gastrocutaneous fistula after laparoscopic sleeve gastrectomy — we performed upper GI endoscopy to all cases first to assess the site , size and cause of fistula . we used stents , clips , sutures and ballon dilatation to close the fistula according to size , site and cause of fistula.if the fistula had no track that was proved by CT with oral & I.V contrast , we used the endoscopic stent. if the fistula had track that was proved by CT with oral & I.V contrast , we used the OVASCO clip , endo suturing or ballon. Combined maneuvers may be used like ballon dilation and clipping or ballon dilatation and suturing if there was distal narrowing.
  Arms: group (2)

SUMMARY:
This study included patients who were admitted to investigators' center to do laparoscopic sleeve gastrectomy and complicated by gastro-cutaneous fistula . Cases were collected in the period from December 2019 to march 2021. The study was approved by the research and Ethics committee of investigators' University .a written informed consent was obtained from all participating patients after explaining to them all the study procedures with its benefits and hazards. the work has been carried out in accordance with the code of ethics of the world medical association ( Declaration of Helsinki ) for studies involving humans .the sample size was calculated using open Epi program using the following data ; confidence interval 95% , power of test 80% , ratio of unexposed/exposed 1, percent of patients with successful management of refractory gastro-cutaneous fistula by surgical intervention 50% and those with successful management by endoscopy 99% , odds ratio 99%, and risk ratio 2 , so the calculated sample size equal 30 patients divided into two equal groups. Group (1) included 15 patients managed by surgical intervention , group (2) included 15 patients managed by endoscopic intervention.

DETAILED DESCRIPTION:
This study included patients who were admitted to investigators' center to do laparoscopic sleeve gastrectomy and complicated by gastro-cutaneous fistula . Cases were collected in the period from December 2019 to march 2021. The study was approved by the research and Ethics committee of investigators' University .a written informed consent was obtained from all participating patients after explaining to them all the study procedures with its benefits and hazards. the work has been carried out in accordance with the code of ethics of the world medical association ( Declaration of Helsinki ) for studies involving humans .the sample size was calculated using open Epi program using the following data ; confidence interval 95% , power of test 80% , ratio of unexposed/exposed 1, percent of patients with successful management of refractory gastro-cutaneous fistula by surgical intervention 50% and those with successful management by endoscopy 99% , odds ratio 99%, and risk ratio 2 , so the calculated sample size equal 30 patients divided into two equal groups. Group (1) included 15 patients managed by surgical intervention , group (2) included 15 patients managed by endoscopic intervention.

Inclusion criteria:

Any patient complicated with gastrocutaneous fistula after laparoscopic sleeve gastrectomy. patients with ASA I & II.

Exclusion criteria:

Any patient complicated with gastrocutaneous fistula after laparoscopic sleeve gastrectomy and managed by conservative measures. Patients with bad general condition ASAIII.

Perioperative measures:

In this randomized control trials , all patients were subjected to the followings: patients were selected by randomization method , Full history taking , Complete physical examination , laboratory investigations ( complete blood picture , liver and kidney functions , coagulation profile ) , radiological investigations ( chest x- ray , ct with oral and i.v contrast to assess if the fistula had track or not ) & patients were subjected to upper GI endoscopy to assess the site , size & cause of fistula .

endoscopic techniques : we performed upper GI endoscopy to all cases first to assess the site , size and cause of fistula . we used stents , clips , sutures and ballon dilatation to close the fistula according to size , site and cause of fistula.if the fistula had no track that was proved by CT with oral & I.V contrast , we used the endoscopic stent. if the fistula had track that was proved by CT with oral & I.V contrast , we used the OVASCO clip , endo suturing or ballon. Combined maneuvers may be used like ballon dilation and clipping or ballon dilatation and suturing if there was distal narrowing.

Follow up after endoscopy and discharge from the hospital:

We examined the patients clinically, made routine laboratory investigations , made follow up ct with oral and i.v contrast & patients were subjected to upper GI endoscopy. The patients were followed up for one week, two weeks and one month, 6months post operatively.

Statistical analysis:

The collected data were analyzed by computer using Statistical Package of Social Services version 22 (SPSS), Data were represented in tables and graphs, Continuous Quantitative variables e.g. age were expressed as the mean ± SD & (range), and categorical qualitative variables were expressed as absolute frequencies (number) & relative frequencies (percentage).

Suitable statistical tests of significance were used after checked for normality. Categorical data were cross tabulated and analyzed by the Chi-square test or Fisher's Exact Test; Continuous data were evaluated by student t- test. The results were considered statistically significant when the significant probability was less than 0.05 (P < 0.05). P-value < 0.001 was considered highly statistically significant (HS), and P-value ≥ 0.05 was considered statistically insignificant (NS).

ELIGIBILITY:
Inclusion Criteria:

* Any patient complicated with gastrocutaneous fistula after laparoscopic sleeve gastrectomy.
* patients with ASA I & II.

Exclusion Criteria:

* Any patient complicated with gastrocutaneous fistula after laparoscopic sleeve gastrectomy and managed by conservative measures.
* Patients with bad general condition ASAIII.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
incidence of recurrence of fistula | within one week after the endoscopy

SECONDARY OUTCOMES:
incidence of side effects of endoscopy | within one month after the endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Said Mohamed Negm, MD, Principal Investigator — ZAGAZIG UNIVERSITY HOSPITALS
Locations (1):
- Zagazig University Hospitals, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Negm S, Mousa B, Shafiq A, Abozaid M, Allah EA, Attia A, AbdelKader T, Farag A. Endoscopic management of refractory leak and gastro-cutaneous fistula after laparoscopic sleeve gastrectomy: a randomized controlled trial. Surg Endosc. 2023 Mar;37(3):2173-2181. doi: 10.1007/s00464-022-09748-z. Epub 2022 Nov 3. PMID 36326931